CLINICAL TRIAL: NCT01693367
Title: A Multi-Center Randomized Controlled Pilot Study of Dynamic Locking Screws 5.0 vs. Standard Locking Screws in Fracture of Distal Femur Treated With Locked Plate Fixation
Brief Title: Dynamic Locking Screws 5.0 vs. Standard Locking Screws in Fracture of Distal Femur Treated With Locked Plate Fixation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The medical device has been withdrawn from the market due to technical issues.
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DLS 5.0
Record Dates: First submitted 2012-09-20; First posted 2012-09-26 (Estimated); Results first posted 2016-07-01 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2016-08

CONDITIONS: Distal Femur Fractures
Keywords: Femoral fracture; Periprosthetic fracture; Fracture fixation, internal; Distal femur fractures; Dynamic Locking Screw; WOMAC
MeSH Terms: conditions — Femoral Fractures, Distal; Femoral Fractures; Periprosthetic Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DLS 5.0 (Dynamic Locking Screws) (Active Comparator): ORIF with DLS 5.0 (Dynamic Locking Screws)
  Interventions: Device: DLS 5.0 (Dynamic locking screws)
- SLS (Standard locking screw) (Active Comparator): ORIF with SLS (Standard locking screw)
  Interventions: Device: SLS (Standard locking screw)

INTERVENTIONS:
Device: DLS 5.0 (Dynamic locking screws) — Open reduction and internal fixation (ORIF) of the distal femur with a large fragment locking plate (LISS, LCP) and DLS 5.0
  Arms: DLS 5.0 (Dynamic Locking Screws)
Device: SLS (Standard locking screw) — Open reduction and internal fixation (ORIF) of the distal femur with a large fragment locking plate (LISS, LCP)and SLS (Standard locking screw)
  Arms: SLS (Standard locking screw)

SUMMARY:
The purpose of this study is to evaluate the performance of Dynamic Locking Screws (DLS) used to stabilize the shaft component of distal femur fractures in comparison to standard locking screws (SLS). The hypothesis is that DLS will lead to better functional outcomes (WOMAC score) due to increased and more symmetrical callus formation and fewer non-unions.

ELIGIBILITY:
Inclusion Criteria:

* 21 years and older
* Closed or open distal femur fracture (AO 33 A1-3, 33 C1-3) including distal femur fractures above a total knee arthroplasty
* Ability to walk independently prior to injury
* Eligible for treatment with ORIF of the distal femur with a large fragment locking plate (LISS, LCP)
* Willing and able to comply with post-operative protocol and return for follow-up.
* Ability to understand the content of the patient information / informed consent form and participate in the clinical investigation
* Signed informed consent

Exclusion Criteria:

* Additional ipsi- or contralateral lower extremity fracture
* Any kind of implant at the ipsilateral proximal femur
* Pre-existing malunion or nonunion of the ipsilateral lower extremity
* Segmental bone defect requiring bone grafting
* More than 4 weeks between injury and surgery
* Pathologic fracture due to a disease other than osteoporosis (eg, tumor, metastasis)
* Polytrauma
* Active malignancy
* Any not medically managed severe systemic disease
* Recent history of substance abuse (ie, recreational drugs, alcohol) that would preclude reliable assessment
* Pregnancy or women planning to conceive within the study period
* Prisoner
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Gardner, MD, Principal Investigator — Washington University School of Medicine; Sean E. Nork, MD, Principal Investigator — University of Washington
Locations (12):
- United States (5):
  - UC Davis Medical Center, Sacramento, California
  - University of Missouri Orthopaedics, Columbia, Missouri
  - Washington University Orthopedics, St Louis, Missouri
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Harborview Medical Center, Seattle, Washington
- Wilhelminenspital, Vienna, Austria
- Germany (3):
  - Charité Berlin, Campus Virchow Klinikum, Berlin
  - Universitätsklinikum des Saarlandes, Homburg
  - BGU Tübingen, Tübingen
- Switzerland (3):
  - Cantonal Hospital Chur, Chur
  - Luzerner Kantonsspital, Lucerne
  - Universitätsspital Zürich, Zurich

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The multicenter international study enrolled patients with distal femur fractures which were either stabilize with a Dynamic Locking Screw or a standard locking screw. The study was stopped due to implant breakages observed after planned implant removals in non-study patients treated with the DLS 5.0mm.
Pre-assignment Details: Five patients signed the informed consent form and were enrolled in the study before it was terminated. Three of the five patients were post-enrollment drop-outs and only two patients completed all study follow-up visits.
Period: Overall Study
Arm/Group | DLS 5.0 (Dynamic Locking Screws) | SLS (Standard Locking Screw)
Started | 2 | 3
Completed | 1 | 1
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Study was stopped
Groups:
- Total: Total of all reporting groups
Arm/Group | DLS 5.0 (Dynamic Locking Screws) | SLS (Standard Locking Screw) | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 68.5 [52 to 85] | 55 [23 to 71] | 60.4 [23 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Switzerland | 0 | 1 | 1
  Germany | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario and McMaster Universities Index (WOMAC)
Description: To assess pain, stiffness, and physical function
Time Frame: 12 months after surgery
Population: Five patients signed the informed consent form and were enrolled in the study before it was terminated. Three of the five patients were post-enrollment drop-outs and only two patients completed all study follow-up visits. No analysis was done. Due to the low number of patients an analysis was not indicated, therefore no results are available.
Arm/Group | DLS 5.0 (Dynamic Locking Screws) | SLS (Standard Locking Screw)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Timed Up-and-go Test (TUG)
Description: The TUG measures the time (in seconds) that it takes for an individual to rise from an armchair (chair seat height = 45 cm / 1.5 feet), walk 3 meters (= 10 feet) to a line drawn on the floor, turn around and return to the chair. The time is measured from a seated position (back against the backrest) with a stopwatch started on the command "ready - go" and stopped when the seated position is reached again.
Time Frame: 12 weeks ± 7 days, 6 months ± 30 days
Population: as for outcome 1
Arm/Group | DLS 5.0 (Dynamic Locking Screws) | SLS (Standard Locking Screw)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quality of Life (EuroQol-5D)
Time Frame: Preoperative, 6 weeks ±7 days, 12 weeks ± 7 days, 6 months ± 30 days, 12 months up to 425 days after surgery
Population: as for outcome 1
Arm/Group | DLS 5.0 (Dynamic Locking Screws) | SLS (Standard Locking Screw)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Range of Motion (ROM)
Description: Assessment of passive ROM of the knee (flexion - extension)
Time Frame: 6 weeks ±7 days, 12 weeks ± 7 days, 6 months ± 30 days, 12 months up to 425 days after surgery
Population: as for outcome 1
Arm/Group | DLS 5.0 (Dynamic Locking Screws) | SLS (Standard Locking Screw)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Full Weight-bearing Status
Description: Assessment of the timepoint when the patient :
  * can bear the whole body weight on the affected leg at single-leg-stance for 3 seconds
  * can walk without walking aid
  * has no intake of analgesics
  * has a pain level experienced at the fracture site during weight bearing over two consecutive measurements with a value of ≤ 3 as measured on a 0-10 numeric rating scale (NRS), where 0 = no pain and 10 = worst pain imaginable
Time Frame: weekly measurement at home
Population: as for outcome 1
Arm/Group | DLS 5.0 (Dynamic Locking Screws) | SLS (Standard Locking Screw)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: WOMAC
Description: To assess pain, stiffness, and physical function
Time Frame: Preoperative, 6 weeks ±7 days, 12 weeks ± 7 days, 6 months ± 30 days, 12 months up to 425 days after surgery
Population: as for outcome 1
Arm/Group | DLS 5.0 (Dynamic Locking Screws) | SLS (Standard Locking Screw)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | DLS 5.0 (Dynamic Locking Screws) | SLS (Standard Locking Screw)
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No